CLINICAL TRIAL: NCT07279298
Title: Effectiveness of Immunization in Preventing Severe Acute Respiratory Infection Associated With Respiratory Syncytial Virus-RSV- in Infants Under 6 Months of Age in Bogotá: a Case-control Study With a Negative Test Design
Brief Title: Effectiveness of Immunization in Preventing Severe Acute Respiratory Infection RSV
Status: Not yet recruiting | Type: Observational
Sponsor: Bogotá District Health Secretariat (Other Government)
Responsible Party: Sponsor
Other Study IDs: SDSCTI20250014
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Syncytial Virus Infections; Severe Acute Respiratory Infection; Bronchiolitis, Viral; Viral Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Bronchiolitis, Viral | interventions — abrysvo; nirsevimab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case (RSV-positive test result): An infant younger than six months of age, resident in Bogotá, hospitalized for severe acute respiratory infection (SARI) and meeting the district operational criteria for SARI, who has a respiratory specimen collected within ≤48 hours of hospital admission (or repeated within 24-48 hours if the first result was negative) that tests positive for Respiratory Syncytial Virus (RSV) by RT-PCR or a validated antigen assay. Only infants born ≥5 weeks after the start of the maternal RSVpreF vaccination campaign are eligible for inclusion.
  Interventions: Biological: RSVpreF vaccine (Abrysvo) and Nirsevimab (Beyfortus) or unexposed
- Control (RSV-negative test result): An infant younger than six months of age, resident in Bogotá, hospitalized for severe acute respiratory infection (SARI) and meeting the same operational criteria as cases, who has a respiratory specimen collected within ≤48 hours of admission (or repeated within 24-48 hours if needed) that tests negative for RSV. Controls may test positive for other respiratory viruses or bacteria. Only infants born ≥5 weeks after the start of the maternal RSVpreF vaccination campaign are eligible.
  Interventions: Biological: RSVpreF vaccine (Abrysvo) and Nirsevimab (Beyfortus) or unexposed

INTERVENTIONS:
Biological: RSVpreF vaccine (Abrysvo) and Nirsevimab (Beyfortus) or unexposed — Maternal vaccination administered between 28 and 36 weeks of gestation and Single-dose monoclonal antibody administered to newborns whose mothers did not receive effective RSVpreF vaccination or unexposed

SUMMARY:
This study aims to evaluate the real-world effectiveness of two preventive immunization strategies against Respiratory Syncytial Virus (RSV)-associated severe acute respiratory infection in infants less than six months of age in Bogotá, Colombia. The strategies include maternal vaccination with RSVpreF administered between 28 and 36 weeks of gestation and neonatal immunization with nirsevimab for infants born to mothers who did not receive RSVpreF during pregnancy. Using a test-negative case-control design embedded in the city's sentinel surveillance system, infants hospitalized for severe respiratory infection will be systematically tested for RSV. Comparative vaccine effectiveness will be estimated to determine the impact of maternal RSV vaccination and neonatal monoclonal antibody immunization on RSV-associated hospitalizations, intensive care admissions, and mortality. The study will generate real-world evidence to inform local and regional public health decisions and guide the implementation of cost-effective hybrid immunization strategies against RSV in middle-income settings.

DETAILED DESCRIPTION:
Respiratory Syncytial Virus (RSV) is a leading cause of hospitalization, morbidity, and mortality among infants, particularly during the first months of life. In 2026, Bogotá will introduce a hybrid immunization strategy combining maternal vaccination with RSVpreF during weeks 28-36 of pregnancy and neonatal immunization with nirsevimab for infants whose mothers were not vaccinated. Despite evidence from clinical trials, real-world comparative effectiveness data for hybrid RSV immunization strategies in Latin America remain limited.

This observational study will employ a prospective test-negative case-control design using the city's sentinel surveillance network for severe respiratory infection. All eligible infants under six months hospitalized for severe acute respiratory infection will undergo laboratory testing for RSV. Cases will be defined as RSV-positive infants, and controls as RSV-negative infants. Exposure to RSVpreF or nirsevimab will be validated through Bogotá's immunization registry.

Primary outcomes include laboratory-confirmed RSV-associated hospitalization, admission to intensive care, and death within the first six months of life. Multilevel logistic regression models adjusted for relevant confounders will be used to estimate vaccine effectiveness. Findings will provide rigorous real-world evidence to support policy decisions, optimize resource allocation, and guide the expansion of hybrid RSV prevention strategies in Colombia and other middle-income countries.

ELIGIBILITY:
Inclusion Criteria:

* Age: Infants younger than 6 months at the time of hospital admission.
* Residence: Maternal residence in Bogotá, Colombia, verified through clinical record, identification document, or health system registry.
* Clinical Condition: Hospitalization due to severe acute respiratory infection (SARI) meeting the district operational definition (presence of fever, cough, and/or signs of respiratory distress, requiring inpatient management).
* Laboratory Testing: Respiratory specimen collected and tested for RSV by RT-PCR or validated antigen test within ≤48 hours of hospital admission, or repeated within 24-48 hours if initial test is negative.
* Exposure Eligibility Window: Infant born ≥5 weeks after the start of the RSVpreF maternal vaccination campaign in Bogotá, ensuring opportunity for maternal immunization.

Exclusion Criteria:

* Prematurity: Infants born at ≤32 weeks of gestation.
* Healthcare-associated respiratory infection: Symptom onset >48 hours after hospital admission for another condition.
* Non-respiratory hospital admission: Primary reason for hospitalization unrelated to respiratory disease (e.g., trauma, elective surgery).
* Vaccination status unverifiable: Inability to confirm maternal RSVpreF vaccination status after reasonable attempts to verify through registry, vaccination card, or prenatal documentation.
* Duplicate episodes: Readmission for the same respiratory episode ≤14 days after discharge (only the first episode will be included).
* Delayed sampling: First respiratory sample obtained >48-72 hours after initial admission to the health system.
* Lethal congenital conditions: Congenital or genetic disorders incompatible with life or that substantially alter the expected clinical course.
* Concurrent interventional study participation: Enrollment in another clinical trial that may affect respiratory outcomes.
* Inability to establish mother-infant linkage due to adoption, loss of parental custody, or absence of biological maternal records.

Ages: 1 Day to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants younger than six months residing in Bogotá, Colombia, hospitalized for severe acute respiratory infection in sentinel hospitals and tested for RSV within 48 hours of admission. The population includes infants exposed to maternal RSVpreF vaccination, neonatal nirsevimab, or neither intervention. Extremely preterm infants (≤32 weeks gestation) and those hospitalized for non-respiratory conditions are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 1097 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Hospitalization for RSV-associated Severe Acute Respiratory Infection | From birth up to 6 months of age (≤180 days of life)
  Proportion of infants hospitalized with laboratory-confirmed Respiratory Syncytial Virus (RSV)-associated severe acute respiratory infection, defined as meeting the district operational criteria for SARI and testing positive for RSV by RT-PCR or validated antigen testing within ≤48 hours of hospital admission. The measure compares the likelihood of RSV-related hospitalization among infants exposed to maternal RSVpreF vaccination, neonatal nirsevimab administration, or no RSV-specific immunization.

CONTACTS AND LOCATIONS:
Overall Officials: Julián Alfredo Fernández Niño, Principal Investigator — Bogotá District Health Secretariat

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coultas JA, Smyth R, Openshaw PJ. Respiratory syncytial virus (RSV): a scourge from infancy to old age. Thorax. 2019 Oct;74(10):986-993. doi: 10.1136/thoraxjnl-2018-212212. Epub 2019 Aug 5. PMID 31383776
- [Background] Mazur NI, Caballero MT, Nunes MC. Severe respiratory syncytial virus infection in children: burden, management, and emerging therapies. Lancet. 2024 Sep 21;404(10458):1143-1156. doi: 10.1016/S0140-6736(24)01716-1. Epub 2024 Sep 9. PMID 39265587
- [Background] Wang X, Li Y, Shi T, Bont LJ, Chu HY, Zar HJ, Wahi-Singh B, Ma Y, Cong B, Sharland E, Riley RD, Deng J, Figueras-Aloy J, Heikkinen T, Jones MH, Liese JG, Markic J, Mejias A, Nunes MC, Resch B, Satav A, Yeo KT, Simoes EAF, Nair H; Respiratory Virus Global Epidemiology Network; RESCEU investigators. Global disease burden of and risk factors for acute lower respiratory infections caused by respiratory syncytial virus in preterm infants and young children in 2019: a systematic review and meta-analysis of aggregated and individual participant data. Lancet. 2024 Mar 30;403(10433):1241-1253. doi: 10.1016/S0140-6736(24)00138-7. Epub 2024 Feb 14. PMID 38367641
- [Background] Everard ML. The relationship between respiratory syncytial virus infections and the development of wheezing and asthma in children. Curr Opin Allergy Clin Immunol. 2006 Feb;6(1):56-61. doi: 10.1097/01.all.0000200506.62048.06. PMID 16505613
- [Background] Mezarina Esquivel, Hugo Antonio, Rojas Medina, Aurea Rosa, Bada Mancilla, Carlos Alfonso, Castañeda Campozano, Ruth Elizabeth, & Carhuancho Aguilar, José Raphael. (2016). Características clínicas y epidemiológicas de la infección respiratoria aguda grave por virus sincitial respiratorio en menores de 5 años. Horizonte Médico (Lima), 16(3), 6-11.
- [Background] Lozano R, Naghavi M, Foreman K, Lim S, Shibuya K, Aboyans V, Abraham J, Adair T, Aggarwal R, Ahn SY, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Barker-Collo S, Bartels DH, Bell ML, Benjamin EJ, Bennett D, Bhalla K, Bikbov B, Bin Abdulhak A, Birbeck G, Blyth F, Bolliger I, Boufous S, Bucello C, Burch M, Burney P, Carapetis J, Chen H, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahodwala N, De Leo D, Degenhardt L, Delossantos A, Denenberg J, Des Jarlais DC, Dharmaratne SD, Dorsey ER, Driscoll T, Duber H, Ebel B, Erwin PJ, Espindola P, Ezzati M, Feigin V, Flaxman AD, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabriel SE, Gakidou E, Gaspari F, Gillum RF, Gonzalez-Medina D, Halasa YA, Haring D, Harrison JE, Havmoeller R, Hay RJ, Hoen B, Hotez PJ, Hoy D, Jacobsen KH, James SL, Jasrasaria R, Jayaraman S, Johns N, Karthikeyan G, Kassebaum N, Keren A, Khoo JP, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lipnick M, Lipshultz SE, Ohno SL, Mabweijano J, MacIntyre MF, Mallinger L, March L, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGrath J, Mensah GA, Merriman TR, Michaud C, Miller M, Miller TR, Mock C, Mocumbi AO, Mokdad AA, Moran A, Mulholland K, Nair MN, Naldi L, Narayan KM, Nasseri K, Norman P, O'Donnell M, Omer SB, Ortblad K, Osborne R, Ozgediz D, Pahari B, Pandian JD, Rivero AP, Padilla RP, Perez-Ruiz F, Perico N, Phillips D, Pierce K, Pope CA 3rd, Porrini E, Pourmalek F, Raju M, Ranganathan D, Rehm JT, Rein DB, Remuzzi G, Rivara FP, Roberts T, De Leon FR, Rosenfeld LC, Rushton L, Sacco RL, Salomon JA, Sampson U, Sanman E, Schwebel DC, Segui-Gomez M, Shepard DS, Singh D, Singleton J, Sliwa K, Smith E, Steer A, Taylor JA, Thomas B, Tleyjeh IM, Towbin JA, Truelsen T, Undurraga EA, Venketasubramanian N, Vijayakumar L, Vos T, Wagner GR, Wang M, Wang W, Watt K, Weinstock MA, Weintraub R, Wilkinson JD, Woolf AD, Wulf S, Yeh PH, Yip P, Zabetian A, Zheng ZJ, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2095-128. doi: 10.1016/S0140-6736(12)61728-0. PMID 23245604
- [Background] Instituto Nacional de Salud (Colombia). Protocolo de vigilancia en salud pública de infección respiratoria aguda. Versión 09 [Internet]. 2024 [citado 2025 Jul 31]. Disponible en: https://doi.org/10.33610/CBNQ7644
- [Background] Hyrkas-Palmu H, Hugg TT, Jaakkola JJK, Ikaheimo TM. The influence of weather and urban environment characteristics on upper respiratory tract infections: a systematic review. Front Public Health. 2025 Feb 10;13:1487125. doi: 10.3389/fpubh.2025.1487125. eCollection 2025. PMID 39995623
- [Background] Deng S, Cong B, Edgoose M, De Wit F, Nair H, Li Y. Risk factors for respiratory syncytial virus-associated acute lower respiratory infection in children under 5 years: An updated systematic review and meta-analysis. Int J Infect Dis. 2024 Sep;146:107125. doi: 10.1016/j.ijid.2024.107125. Epub 2024 Jun 28. PMID 38945430
- [Background] Galvis, Clara Esperanza, Troncoso, Gloria, Agudelo-Pérez, Sergio, Romero, Héctor, Parra Buitrago, Andrea, & Gutiérrez, Iván Felipe. (2024). Consenso de expertos sobre las recomendaciones de profilaxis con palivizumab para el Virus Sincitial Respiratorio en niños en Colombia. Infectio, 28(3), 180-191. Epub September 12, 2024.https://doi.org/10.22354/24223794.1189
- [Background] Novoa Pizarro JM, Lindemann Tappert BC, Luchsinger Farias VR, Vargas Munita SL. [Prevention of respiratory syncytial virus infection in infants. What has been done and where are we today?]. Andes Pediatr. 2023 Dec;94(6):672-680. doi: 10.32641/andespediatr.v94i6.4861. Spanish. PMID 38329302
- [Background] Hammitt LL, Dagan R, Yuan Y, Baca Cots M, Bosheva M, Madhi SA, Muller WJ, Zar HJ, Brooks D, Grenham A, Wahlby Hamren U, Mankad VS, Ren P, Takas T, Abram ME, Leach A, Griffin MP, Villafana T; MELODY Study Group. Nirsevimab for Prevention of RSV in Healthy Late-Preterm and Term Infants. N Engl J Med. 2022 Mar 3;386(9):837-846. doi: 10.1056/NEJMoa2110275. PMID 35235726
- [Background] Kampmann, B., et al. (2023).
- [Background] Torres JP, Saure D, Goic M, Thraves C, Pacheco J, Burgos J, Trigo N, Del Solar F, Neira I, Diaz G, O'Ryan M, Basso LJ. Effectiveness and impact of nirsevimab in Chile during the first season of a national immunisation strategy against RSV (NIRSE-CL): a retrospective observational study. Lancet Infect Dis. 2025 Nov;25(11):1189-1198. doi: 10.1016/S1473-3099(25)00233-6. Epub 2025 Jun 10. PMID 40513593
- [Background] Perez Marc G, Vizzotti C, Fell DB, Di Nunzio L, Olszevicki S, Mankiewicz SW, Braem V, Rearte R, Atwell JE, Bianchi A, Fuentes N, Zadoff R, Vecchio G, Gabriela Abalos M, Fan R, Del Carmen Morales G, Gessner BD, Jodar L, Libster R, Rearte A; BERNI study working group. Real-world effectiveness of RSVpreF vaccination during pregnancy against RSV-associated lower respiratory tract disease leading to hospitalisation in infants during the 2024 RSV season in Argentina (BERNI study): a multicentre, retrospective, test-negative, case-control study. Lancet Infect Dis. 2025 Sep;25(9):1044-1054. doi: 10.1016/S1473-3099(25)00156-2. Epub 2025 May 5. PMID 40339585
- See also: cost analysis — https://www.saludcapital.gov.co/DSP/Sincitial/Anx_3_analisis_costo_efec.pdf
- See also: Boletin epidemuiologico — https://www.ins.gov.co/buscador-eventos/Paginas/Vista-Boletin-Epidemilogico.aspx